CLINICAL TRIAL: NCT04262713
Title: Evaluation of Predictive Factors for Ruptures of Meije Duo ™ Size 1 and 2 Femoral Stems in Hip Replacement Surgery
Acronym: MEIJE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, SMARMOR, orthopedic surgeon, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ID RCB : 2018-A02841-54
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hip Arthropathy Associated With Other Conditions
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients implanted with Meije duo stem size 1 or 2 (Other): Among this arm, patients that meet criteria ( weight>
  60kg and / or a long neck / varus and / or a DEVANE score ≥ 4 ) will perform hip X ray
  Interventions: Other: Radiographs

INTERVENTIONS:
Other: Radiographs — Radiographs of the implanted hip with Meije duo size1 or 2 are performed in eligible patients ( Weigh>60, Long neck stem, Varus; DEVANE score ≥ 4)

SUMMARY:
A normative development concerning the mechanical resistance tests of the the femoral stems led to contraindicate, in September 2014, to implant Meije Duo ™ femoral stems size 1 or 2 in patients weighing more than 60 kg due to an assumed risk of femoral stem breakage.

This contraindication is based on standardized mechanical tests which may have not taken into account the changes in patient weight that may occur after the intervention.

To date, investigators have not been aware of any Meije Duo ™ size 1/2 brakeage in our patients implanted with this type of prosthesis regardless of their weights before 2014. However, it is possible that some of them have had a prostheses failure and consulted another hospital. In the absence of a clinical study on this problem, investigators decided to set up a health care assessment study collecting retrospective and prospective information from our patients.

DETAILED DESCRIPTION:
First, patients with Meije Duo ™sizes 1 or 2, who had surgery from 2007 to 2014, will be preselected on medical records.

The information notice will be sent to them by post. A period of reflection will be respected before contacting the patient to answer their questions concerning the research and its progress and obtain their oral consent to participate in the study.

After obtaining consent, investigators will enter the retrospective data collected in the medical and prospective file collected during this call.

Patients with at least one of the following criteria: weight> 60 kg and / or long neck / varus and / or DEVANE score ≥ 4, will be selected to have a hip X-ray which will be specially scheduled for the study.

This examination will tell us about the state of the prosthesis and of the underlying bone (broken stem, loosening of the implant, bone fracture, dislocation, border, etc.

It can be performed in our radiology department of the Diaconesses Croix Saint Simon hospital group or in another radiological center chosen by the patient if the latter cannot come to our hospital. In this case, a prescription for a hip X-ray will be sent to him by post to his current address as well as an information letter intended for the radiology office.

The patients who will be included in the study are implanted with Meije Duo ™ 1 and 2 between 2007 to 2014 and will all have a minimum follow-up of 4 years from the date of implantation. The maximum number of rupture complications is observed between the fourth and the eleventh year after fitting the prosthesis. All participants will therefore have a minimum of hindsight required for the evaluation of stem breaks. All of our patients will be contacted by telephone during the study period in chronological order of their previous management for obtaining consent, prospective data and for scheduling the hip radiography according to the criteria mentioned above.

ELIGIBILITY:
Inclusion Criteria:

An x-ray of the hip concerned will be performed on all consenting patients, having at least one criterion of the following three during their medical history since the implantation of the hip prosthesis.

* Weight> 60 kg
* DEVANE score ≥ 4
* Long neck / varus

Exclusion Criteria:

* The patient expresses his opposition to the use of his personal data
* Patients (<18 years old)
* Patients unable or out of state to express their consent
* Patient unable to speak French
* Patient with memory impairment or cognitive impairment
* Patient not affiliated to a social security or equivalent health coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Pourcentage of participants who had stem (Meije DuoTM size 1 or 2) breakage occured between implantation and the study follow-up call phone. | Up to 4 weeks, starting from the call phone (patient consent)
  The number of stem breakage that occured since prostheses implantation will be collected by asking every participant during the follow-up call phone and performing hip xray to eligible ones (see above)

SECONDARY OUTCOMES:
Pourcentage of participants who had other prostheses failures (loosening of the prosthesis, femoral fracture, dislocation) | Up to 4 weeks, starting from the call phone (patient consent)
  The number of prostheses failures that occured since the implantation will be collected by asking every participant during the follow-up call phone and by performing hip xray to eligible ones (see above)
The change of physical activity in participants from baseline (prostheses implantation) to study call-phone point time. | Change from baseline Devane score at postoperative 4 years
  With DEVANE questionnaire, investigator will assess physical activity of participants
The change of the weight and the body mass index (BMI) of the patients after the implantation of Meije DuoTM rods size 1 or 2 | Change from baseline weight and BMI at postoperative 4 years
  Preoperative weight and BMI of particpantS will be collected from the medical file and postopeartive weight and BMI during follow up call phone

CONTACTS AND LOCATIONS:
Overall Officials: Simon MARMOR, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (4):
- France (4):
  - Groupe Hospitalier Diaconesses Croix saint Simon, Paris
  - Orthopedic department, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region
  - Groupe Hospitalier Dianconesses croix saint Simon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wroblewski BM, Siney PD, Fleming PA. Increasing patients' body mass. Are the criteria for testing stemmed femoral components in total hip arthroplasty still valid? Proc Inst Mech Eng H. 2007 Nov;221(8):959-61. doi: 10.1243/09544119JEIM305. PMID 18161256
- [Background] Silva M, Shepherd EF, Jackson WO, Dorey FJ, Schmalzried TP. Average patient walking activity approaches 2 million cycles per year: pedometers under-record walking activity. J Arthroplasty. 2002 Sep;17(6):693-7. doi: 10.1054/arth.2002.32699. PMID 12216021
- [Result] Westerman AP, Moor AR, Stone MH, Stewart TD. Hip stem fatigue: : The implications of increasing patient mass. Proc Inst Mech Eng H. 2018 May;232(5):520-530. doi: 10.1177/0954411918767200. Epub 2018 Apr 2. PMID 29608134